CLINICAL TRIAL: NCT03507764
Title: Evaluation of a Treadmill Workstation in an Emergency Dispatch Center. A Randomized Controlled Trial.
Brief Title: Evaluation of a Treadmill Workstation in an Emergency Dispatch Center
Acronym: Marche_15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Marche pour le 15
Record Dates: First submitted 2018-02-12; First posted 2018-04-25 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2019-08

CONDITIONS: Work-Related Condition
Keywords: Treadmills; Exercise; Number of steps; Dispatchers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): During the randomized study phase (6 months),subjects will perform their usual activity without access to the treadmill workstation in the dispatch center.
  After six months, all subjects will continue to be assessed with free access to the treadmill workstation at the workplace.
- Experimental Group (Experimental): During the randomized study phase, subjects will have an open access to the treadmill workstation with the indication to use it for at least one hour (continuous or split) on working days.
  After six months, all subjects will continue to be assessed with free access to the treadmill workstation.
  Interventions: Other: Use of the treadmill workstation at work

INTERVENTIONS:
Other: Use of the treadmill workstation at work — During the randomized study phase, provision of the treadmill workstation with the recommendation to use it for at least one hour (continuous or split) during each of the working shifts.
  After six months, all subjects will use treadmill without restrictions or conditions.
  Arms: Experimental Group

SUMMARY:
The principal objective of this study is to determine if the provision of a treadmill workstation in an emergency medical services (EMS) dispatch center increases the number of steps that participants make daily within 6 months compared to the usual working conditions.

The investigators hypothesized that the provision of a treadmill workstation with a slow walking could increase the number of daily steps and decrease days of leave, musculoskeletal disorders without decreasing the dispatch quality.

DETAILED DESCRIPTION:
Sedentariness, measured by the daily duration of time spent seated is a cardiovascular risk factor, chronic pathologies (cancer, musculoskeletal pain) and mortality.

The employees who remain seated from 8 to 11 hours per day have an increase risk of death within 3 years (15%). This increase reaches 40% for more than 11 hours a day.

The restoration of a daily moderate physical activity from 60 to 75 minutes could permit to eliminate this increased risk.

Interventions in workplace to limit sitting are associated with a metabolic benefit, but also with a reduction in musculoskeletal problems and fatigue.

The role of dispatchers is to initiate the medical record by determining the severity of the call and take rapid and adequate decision.

They are seated behind their desks from 8 to 11 hours in a busy and stressful environment.

Many dispatchers are complaining of musculoskeletal disorders and weight gain. An internal study conducted between between 2012 and 2016 showed an increase in long-term pain, irritability and sleep disorders. Overall, 65% of the respondents reported that they were tired at work and had less empathy.

The use of workstations with low-speed treadmills were assessed to allow physical activity at work.

A recent review concluded that their use reduced the time that the employees spent seated, stress and improved energy expenditure, as well as different biological and physical parameters (weight loss, lipid determination, glycaemia). This study did not reveal any alterations in performance at work.

The investigators assume that the establishment of a position allowing slow walk during dispatch call would increase the number of steps made by dispatchers on a daily basis and reduce the number of days of leave and musculoskeletal disorders, without impairing the quality of call pick-up.

ELIGIBILITY:
Inclusion Criteria:

* Dispatchers working in Emergency Medical Service

Exclusion Criteria:

* Pregnant women
* Inability to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Difference of number of steps at 0 and 6 months | 0 and 6 months
  Number of daily steps measured by actimetry (including all walking activities measured over a day).
  Measurements will be done with actimetry during one week before the randomization and at 6 months

SECONDARY OUTCOMES:
Evaluation of Quality of life | 0, 6 and 12 months
  Assessment of quality of life with the validated Short Form Health Survey assessment SF-36
Evaluation of Anxiety and depression | 0, 6 and 12 months
  Assessment of anxiety depression with the validated Hospital Anxiety and Depression Score.
  This questionnaire helps your physician to know how the patient is feeling.
Change in blood pressure | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Assessment of blood pressure every month
Change in heart rate | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Assessment of heart rate every month
Change in Weight | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Assessment of weight every month
Assessment of musculoskeletal disorders | 0, 6 and 12 months
  Assessment with the validated Standardised Nordic Questionnaire
Evaluation of non-attendance at work | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Number of workdays not realised during the month
Job performance evaluation | 0, 6 and 12 months
  Assessment with the Likert scale (7-points scale) Level of Performance - 7 point 0 - Not at all performant
  1. - Low performant
  2. - Slightly performant
  3. - Neutral
  4. - Moderately performant
  5. - Very performant
  6. - Extremely performant
Work satisfaction evaluation | 0, 6 and 12 months
  Assessment with the Utrecht Work Engagement Scale (7-points scale). Level of Satisfaction - 7 point 0 - Completely dissatisfied
  1. - Mostly dissatisfied
  2. - Somewhat dissatisfied
  3. - neither satisfied or dissatisfied
  4. - Somewhat satisfied
  5. - Mostly satisfied
  6. - Completely satisfied
Assessment of sleep quality | 0, 6 and 12 months
  Assessment with the Pittsburgh Quality Index survey
Evaluation of tobacco consumption | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Mean of packs of smoked cigarettes during the week before the evaluation. This evaluation is based on a declared and quantitative consumption.
Evaluation of pickup calls quality | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Calls are evaluated according to the following criteria:
  * Presentation of the volunteer at the picked up of the call
  * Audio quality
  * Listening of the patient request
  * Empathy
  * Relevance of the call sort
  * Management of the end of communication
  * Call duration
Walking period during a working day | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months
  Evaluation of walking time on the treadmill with the integrated software

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Debaty, MD, PhD, Principal Investigator — CHU Grenoble Alpes, SAMU38
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No